CLINICAL TRIAL: NCT04682496
Title: Evaluation of the Influence of Ultrasound Probe Pressure on the Intratendon Doppler Signal in Patellar Tendinopathy
Brief Title: Ultrasound Probe Pressure on the Intratendon Doppler Signal in Patellar Tendinopathy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cardenal Herrera University (Other)
Responsible Party: Principal Investigator, SERGIO MONTERO NAVARRO, Principal Investigator, Cardenal Herrera University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CEI20/073
Record Dates: First submitted 2020-12-09; First posted 2020-12-23 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2023-02

CONDITIONS: Patellar Tendinitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- intratendon vascularization (Experimental): Intratendon vascularization will be quantified using a proprietary methodology using ImageJ 1.47v image analysis software, determining the different variables related to the Doppler signal within an intratendon region of interest.
  Interventions: Procedure: Intratendon vascularization

INTERVENTIONS:
Procedure: Intratendon vascularization — Ultrasonic exploration by power-Doppler of the intratratendon vascularization, making longitudinal cuts of the patellar tendon and with previously pre-established Doppler optimization parameters for all patients. The optimization parameters of the power-Doppler signal will be set at a Doppler frequency of 6.7 MHz, pulse repetition frequency (PRF) of 0.7 kHz. The lowest wall filter and a standardized gain just below the level that produces random noise will be applied. This examination will be repeated several times with different probe pressures, which will be quantitatively adjusted through the force sensor and maintained with the articulated arm. A 4-second static video will be recorded of the longitudinal section that presents a higher Doppler signal in each of the scans at different probe pressures.

SUMMARY:
In the sports field, patellar tendinopathy is, as a pathology, one of the main concerns for athletes, both because of its incidence and because of the difficulty involved in their recovery. At the ultrasound level, tendinopathies can be divided, depending on the presence or absence of an intratendon Doppler signal, into hypervascular or hypovascular tendinopathy. Its classification is, today and clinically speaking, merely qualitative through the observation of the explorer. The ultrasound evaluation is carried out through a probe that is placed on the patient's skin, the procedure to be followed to obtain a vascular image is merely operator-dependent, that is, the position of the probe, the pressure exerted on the skin or even ultrasound optimization parameters can drastically modify the results.

Due to high pressure on the probe, the intratendon Doppler signal may be diminished in the quantitative variables of area, number of signals, pixel intensity, perimeter, solidity, perfusion index, circularity, major and minor diameter.

From a certain pressure on the probe, the intratendon Doppler signal can be drastically altered.

This study will try to evaluate the influence of the pressure exerted by the examiner with the probe on the quantitative variables of the intratendon Doppler signal in patellar tendinopathy.

To carry out the study, a single group with patellar tendinopathy will be established. Ultrasound evaluations with Doppler mode will be performed on the tendon using different probe pressures, monitoring the applied force and recording the images obtained for later analysis.

ELIGIBILITY:
Inclusion Criteria:

* Acceptance of participation in the study.
* Diagnosis of patellar tendinopathy with the presence of an intratendon Doppler signal.
* Subjects between the ages of 18 and 65.

Exclusion Criteria:

* Present some type of surgical intervention in the region to be explored that could alter in some way the ultrasound evaluation.
* Refer vascular pathology or the intake of medication that may alter blood flow or density.
* Having been treated with sclerosing techniques that can alter the perfusion or vascular resistance of the tendon tissue.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2020-12-18 (Actual); Primary Completion 2022-08-30 (Actual); Study Completion 2023-02-07 (Actual)

PRIMARY OUTCOMES:
number of signals (n) | during intervention
  number of intratendon doppler signals (unit)
Average pixel intensity (0-255 Units on a scale) | during intervention
  average pixel color intensity (0-255 Units on a scale)
Area (mm^2) | during intervention
  intratendon Doppler signal area (mm^2)
Perimeter (mm) | during intervention
  perimeter of the intratendon Doopler signal (mm)
major diameter (mm) | during intervention
  major diameter of the intratendon Doppler signal (mm)
minor diameter (mm) | during intervention
  minor diameter of the intratendon Doppler signal (mm)
Circularity | during intervention
  measure of roundness or circularity, area-to perimeter ratio. (0-1 Units on a scale)
Solidity | during intervention
  measures the density of an object (0-1 Units on a scale)
Resistance index | during intervention
  resistance index of intratendon Doppler signals (0-1 Units on a scale)
Force | during intervention
  force applied by the probe on the knee during the scan (N)

SECONDARY OUTCOMES:
Age (years) | Post-intervention
  subject's age (years)
Sex (female or male) | post-intervention
  subject's sex (female or male)
Time of evolution (months) | months
  time since the patient had the first symptoms (months)
Dominance | post-intervention
  Dominant leg (right-left)
Pain location | Immediately pre-intervention
  Location of pain in the patellar tendon (lower pole of the patella-body of the tendon-insertion in the anterior tuberosity of the tibia)
Victorian Institute of Sport Assessment-Patella (VISA-P) | Immediately pre-intervention
  Knee pain and function rating scale (0-100 Units on a scale). The maximum score possible is 100 points and represents an asymptomatic athlete who can fully engage in sports. The theoretical minimum is 0 point. The test is carried out just before the intervention to relate the results of the Doppler quantification with the severity of the pain.
hours of training (hours) | Immediately pre-intervention
  Current training hours per week (hours). This question is asked just before the intervention in order to relate the results of the Doppler quantification with the hours of training performed
Time without training (months) | Immediately pre-intervention
  time without training (months). This question is asked just before the intervention.

CONTACTS AND LOCATIONS:
Locations (1):
- Ceu Cardenal Herrera University, Elche, Alicante, Spain

REFERENCES:
- [Background] Hernandez-Sanchez S, Hidalgo MD, Gomez A. Cross-cultural adaptation of VISA-P score for patellar tendinopathy in Spanish population. J Orthop Sports Phys Ther. 2011 Aug;41(8):581-91. doi: 10.2519/jospt.2011.3613. Epub 2011 Jul 12. PMID 21765223
- [Background] Dhyani M, Roll SC, Gilbertson MW, Orlowski M, Anvari A, Li Q, Anthony B, Samir AE. A pilot study to precisely quantify forces applied by sonographers while scanning: A step toward reducing ergonomic injury. Work. 2017;58(2):241-247. doi: 10.3233/WOR-172611. PMID 28922185
- [Background] Malliaras P, Chan O, Simran G, Martinez de Albornoz P, Morrissey D, Maffulli N. Doppler ultrasound signal in Achilles tendinopathy reduces immediately after activity. Int J Sports Med. 2012 Jun;33(6):480-4. doi: 10.1055/s-0032-1304636. Epub 2012 Apr 12. PMID 22499574
- [Background] Boesen AP, Boesen MI, Torp-Pedersen S, Christensen R, Boesen L, Holmich P, Nielsen MB, Koenig MJ, Hartkopp A, Ellegaard K, Bliddal H, Langberg H. Associations between abnormal ultrasound color Doppler measures and tendon pain symptoms in badminton players during a season: a prospective cohort study. Am J Sports Med. 2012 Mar;40(3):548-55. doi: 10.1177/0363546511435478. Epub 2012 Feb 9. PMID 22328709
- See also: The University CEU-Cardenal Herrera is th first private university in the Valencian Community. It belongs to the Foundation San Pablo - CEU and is the leading educational organization in Spain with three Universities all over Spain — http://www.uchceu.es

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2020-12-12): https://cdn.clinicaltrials.gov/large-docs/96/NCT04682496/Prot_SAP_ICF_000.pdf